CLINICAL TRIAL: NCT05559827
Title: Randomized Prospective Trial Evaluating the Efficacy of the antiCD38 Monoclonal Antibody Isatuximab in the Treatment of PCRA by Major ABO Mismatch After Allogeneic Hematopoietic Stem Cell Transplantation
Brief Title: Efficacy of the antiCD38 Monoclonal Antibody Isatuximab in the Treatment of PCRA by Major ABO Mismatch After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: ErythroSIM
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200067
Record Dates: First submitted 2022-09-14; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Immunological Pure Red Cell Aplasia
MeSH Terms: interventions — isatuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isatuximab arm (Experimental): Isatuximab treatment at a dose of 10 mg/kg by intravenous route. The first injection of isatuximab will be performed at randomization (month 6 +/- 2 days). A second injection may be performed at day 15 if the reticulocytes <10 G / L, and a third at day 29 if reticulocytes <10 G / L. Patients will be assessed on day 1, day 15, day 29, day 45, 2 months, 3 months, 6 months and 9 months after randomization.
  Interventions: Drug: Isatuximab
- comparator arm (No Intervention): No treatment, supportive care will be allowed.

INTERVENTIONS:
Drug: Isatuximab — Isatuximab treatment at a dose of 10 mg/kg by intravenous route. The first injection of isatuximab will be performed at randomization (month 6 +/- 2 days). A second injection may be performed at day 15 if the reticulocytes <10 G / L, and a third at day 29 if reticulocytes <10 G / L. Patients will be assessed on day 1, day 15, day 29, day 45, 2 months, 3 months, 6 months and 9 months after randomization.
  Arms: Isatuximab arm

SUMMARY:
A quarter of allogeneic hematopoietic stem cell transplantation are performed in a situation of major ABO mismatch exposing patients to the risk of immunological pure red cell aplasia (PRCA) after transplant. PCRA after transplant is defined as anemia with low reticulocytes count (under 10 G/L) after day 60 despite good leucocytes and platelet engraftment, full donor chimerism, associated with the persistence of recipients hemagglutinins (anti-A or anti-B antibodies). Bone marrow evaluation when performed show erythroid hypoplasia. Red blood cells transfusions are necessary every two weeks until remission leading to impaired quality of life (anemia, repeated hospitalization), iron overload, and need for iron chelation therapy. Treatments currently used are inefficient (anti CD20 monoclonal antibodies, EPO, steroids, plasma exchanges, proteasome inhibitors) or at risk of severe acute GVHD (donor lymphocytes infusion). PRCA has been demonstrated to be associated with the persistence of recipient's plasma cells.

Anti-CD38 monoclonal antibodies which targets plasma cells secreting hemagglutinins responsible of PCRA are a promising treatment: 6 cases reported in the literature support a rapid and sustain efficacy but a prospective randomized evaluation of its efficacy and safety in this context is necessary.

The main objective of the study is to assess the efficacy of the treatment of PRCA by isatuximab after allogeneic hematopoietic stem cell transplant compared to supportive care only control group (reduction in PRCA resolution time in days)

ELIGIBILITY:
Inclusion Criteria:

* Aged 15 years or older
* Having receiving an allogeneic hematopoietic stem cell transplantation in condition of major ABO mismatch
* PCRA defined by persistent red blood cell transfusion dependence at day 60 post-transplant with reticulocytes count under 10 G/L despite full donor chimerism and a good leucocytes (>1 G/L) and platelet (>50G/L) recovery
* No relapse or progression of underlying disease
* Contraception methods must be prescribed during all the duration of the research and using effective contraceptive methods during treatment for women of childbearing age (continue abstinence from heterosexual intercourse is accepted) and for man during the study treatment period and for at least 5 months after the last dose of study treatment and refrain from donating sperm during this period
* With health insurance coverage
* Having signed a written informed consent (2 parents for patients aged less than 18)

Exclusion Criteria:

* Aged < 15 years
* Relapse of underlying disease
* Leucocyte chimerism < 95%
* PRCA related to Parvovirus B19 infection (positive blood PCR)
* Known to be HIV+ or to have hepatitis A, B, or C active infection
* Active tuberculosis
* Pregnancy (βHCG positive) or breast-feeding.
* Patient receiving recombinant human erythropoietin.
* Patient receiving proteasome inhibitor (Bortezomib for example).
* Patient receiving thrombopoietin receptor agonists (ARTPO).
* Patient receiving plasma or plasmapheresis exchanges after transplant.
* Planned to receive any investigational drug within 14 days or 5 half-lives of the investigational drug, whichever is longer.
* Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose excessive risk to the patient or may interfere with compliance or interpretation of the study results.
* Hypersensitivity to the active substance or history of intolerance to steroids, mannitol, pregelatinized starch, sodium stearyl fumarate, histidine (as base and hydrochloride salt), arginine, hydrochloride, poloxamer 188, sucrose or any of the other components of study therapy that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
* Who have any debilitating medical or psychiatric illness
* Under tutorship or curatorship
* Who not understand informed consent for an optimal treatment and follow-up

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
time interval between randomization (corresponding to the M6 post-transplant) and resolution of PRCA (date of resolution of reticulocytopenia) treated or not by the anti-CD 38 monoclonal antibody isatuximab | 9 months post randomization

SECONDARY OUTCOMES:
Number of red blood cell transfusions after randomization | from randomization through study completion, an average of 9 months after randomization
Ferritin levels | at month 6 post-transplant
Ferritin levels | at month 9 post-transplant
Ferritin levels | at month 15 post-transplant
Adverse events (CTC-AE grade ≥ 2) | up to 13 months post transplant
Quality of life questionnaire (EORTC QLQ-C30- v3) | at day 60
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life questionnaire (EORTC QLQ-C30- v3) | at day 100
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life questionnaire (EORTC QLQ-C30- v3) | at 6 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life questionnaire (EORTC QLQ-C30- v3) | at 9 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life questionnaire (EORTC QLQ-C30- v3) | at 12 months
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Quality of life questionnaire (EORTC QLQ-C30- v3) | at 15 months post-transplant
  Quality of life evaluated using questionnaire "European Organization for Research and Treatment of Cancer Quality of Life Questionnaire" (EORTC QLQ-C30- v3). The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level. A high score for a functional scale represents a high/healthy level of functioning. A high score for the global health status/ QoL represents a high QoL and a high score for a symptom scale/item represents a high level of symptomatology/problems.
Spontaneous resolution of PRCA between day 60 and 6 months post-transplant | at 6 months post-transplant
Antibody level (anti A and/or anti B titers) | at day 60 post transplant
Antibody level (anti A and/or anti B titers) | at day 100 post transplant
Antibody level (anti A and/or anti B titers) | at day 15 post randomization
Antibody level (anti A and/or anti B titers) | at day 29 post randomization
Antibody level (anti A and/or anti B titers) | at day 45 post randomization
Antibody level (anti A and/or anti B titers) | at month 3 post randomization
Antibody level (anti A and/or anti B titers) | at month 6 post-randomization
Antibody level (anti A and/or anti B titers) | at month 9 post-randomization
Number of days of hospitalization | up to 9 months post ranomization
Number of days of transfusions support | up to 9 months post randomization
Number of days of chelation treatments | up to 9 months post randomization

IPD SHARING:
Plan to Share IPD: Undecided